CLINICAL TRIAL: NCT04787094
Title: The Effect of Yoga and Stabilization Exercises on Pain, Functional Status, Metabolic Capacity and Sleep Quality in Individuals With Chronic Low Back Pain: A Randomized, Crossover Study.
Brief Title: The Effect of Yoga and Stabilization Exercises in Individuals With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozlem Ulger, Professor, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KA-20031
Record Dates: First submitted 2021-02-08; First posted 2021-03-08 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Low Back Pain
Keywords: spinal stabilization exercise; yoga; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): The sessions will begin with breathing exercises in standing, sitting, supine and prone positions, and these exercises will be applied for about 10 minutes. After the breathing exercises, the sudden relaxation technique, which will take 2-3 minutes, firstly contracting the whole body from the feet to the head and then completely relaxing it.
  Interventions: Other: Yoga
- Spinal Stabilization Exercise Group (Experimental): Spinal stabilization exercises will be applied to the individuals in this group for 8 weeks / 2 days a week, approximately 50-60 minutes a day under the supervision of a physiotherapist.
  Spinal stabilization exercises will be progressed in 3 phases by gradually increasing the difficulty.
  Interventions: Other: Spinal Stabilization Exercise

INTERVENTIONS:
Other: Yoga — Yoga
  Arms: Yoga Group
Other: Spinal Stabilization Exercise — Spinal Stabilization Exercise
  Arms: Spinal Stabilization Exercise Group

SUMMARY:
Although exercise has been shown to be effective in low back pain in the literature, there is no conclusion about which exercise is superior to the other. Although there are studies showing positive effects of spinal stabilization exercises and yoga approach on pain level, disability level and quality of life in patients with chronic low back pain, studies evaluating the effectiveness in many other aspects are insufficient. Therefore, this study aimed to investigate the effects of spinal stabilization and yoga exercises on pain, functional status, metabolic capacity, kinesophobia and sleep quality in patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific low back pain diagnosis
* Having pain that persists for at least 12 weeks
* 25-65 age range

Exclusion Criteria:

* Scoliosis with a cobb angle of more than 20º
* History of previous surgery for the lumbal region
* Having an additional diagnosis such as spondylolisthesis, spinal stenosis, spondylolysis
* Presence of neurological deficits
* Metastatic state presence
* Presence of neurological deficits due to diabetes
* Presence of metabolic problems such as thyroid, hypertension, coronary artery disease
* The presence of inflammatory problems involving the spine

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 15 minutes, through study completion, an average of 8 weeks, Change from pain intensity
  Pain intensity of participants will be evaluated with visual analog scale (VAS). Paricipants asked to mark the intensity of pain on a 10 cm long line, explaining that the leftmost of the line does not have pain, that the pain increases while moving to the right, and that the pain is unbearable on the far right. VAS scored between 0-10 cm.
Disability Severity | 5 minutes, through study completion, an average of 8 weeks, Change from disability
  Patient's pain related functional status will be measured by Oswestry Disability Index. The scale is considered the 'gold standard' of low back functional outcome tools. This scale contain questions related to functional activities of pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling. Interpretation of scale are 0% to 20% for minimal disability, 21% to 40% for moderate disability, 41 % to 60 % for severe disability 61% to 80 % for crippled and 81 % to 100 % Bed-bound. The Oswestry Disability Index is scored between 0-50 points. An increase in score indicates a poor result.
  Patient's back-related functional performance will be evaluated with Back Performance Scale. Each question is scored between 0 and 3. The total score recorded. The Back Performance Scale test is scored between 0-15 points. An increase in score indicates a poor result.
Funcitonal Performance | 10 minutes, through study completion, an average of 8 weeks, Change from Functional status and performance
  Patient's back-related functional performance will be evaluated with Back Performance Scale. Each question is scored between 0 and 3. The total score recorded. The Back Performance Scale test is scored between 0-15 points. An increase in score indicates a poor result.

SECONDARY OUTCOMES:
Deep muscle activation | 5 minutes, through study completion, an average of 8 weeks, Change from deep muscle activation
  To evaluate the transversus abdominis muscle activation, the stabilizer biofeedback device is placed under the abdomen, just below the spina iliaca anterior superior, while the patient is in the prone position. The cuff of the device is inflated to 70 mmHg, the patient is asked to breathe and pull the abdomen up and in while exhaling, but the patient is warned not to make pelvis and spine movement. In the meantime, how much the pressure has changed is observed from the stabilizer device. In the test, the average of 3 repetitions will be recorded. With successful measurement, the pressure is expected to drop between 6 and 10 mm-Hg.
Kinesiophobia | 5 minutes, through study completion, an average of 8 weeks, Change from kinesiophobia
  Fear-Avoidance-Beliefs Questionnaire will be applied to evaluate kinesiophobia which is fear of movement due to low back pain. This questionnaire has 2 sub-sections related to physical activity and work. There are 4 questions scored in the physical activity section and 7 questions in the work section. 0-6 points are obtained for each question. The total score will be recorded. Physical Activity sub-section scored between 0-24 points. Work sub-sections scored between 0-42 points. The higher the score, the higher the kinesiophobia.
Sleep quality | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline sleep quality
  The Pittsburg Sleep Quality Index will be used to evaluate sleep quality. This questionnaire evaluates sleep quality and disturbance over the past month. The scale consists of 7 subcomponents: Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disturbances, Use of Sleeping Medication, and Daytime Dysfunction. Each component is scored between 0-3 points. The total score of the 7 components gives the total score of the scale. The total score ranges from 0-21. A total score greater than 5 indicates "poor sleep quality".
Metabolic Capacity | 15 minutes, through study completion, an average of 8 weeks, Change from Baseline metabolic capacity.
  Metabolic capacity evaluation will be performed according to 6 Minute Walk Test. Individuals are asked to walk as fast as possible for 6 minutes without running on the 30 m long corridor. The test is started, the number of rounds is recorded while the patient is walking. Heart rate, blood pressure, oxygen saturation and respiratory frequency will be evaluated and recorded at first, at the end of the test and one minute after. Walking distance is recorded in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ülger, Prof, Principal Investigator — Hacettepe University
Locations (1):
- Özlem Ülger, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No.